CLINICAL TRIAL: NCT01452971
Title: A Study of the Interaction Between Tumor Susceptibility Gene GNMT and Lung Cancer
Brief Title: A Study of the Interaction Between Tumor Susceptibility Gene Glycine N-methyltransferase (GNMT) and Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DMR99-IRB-196
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Lung Cancer
Keywords: tumor susceptibility gene; glycine N-methyltransferase (GNMT); polycyclic aromatic hydrocarbons (PAHs); lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Environmental carcinogens such as polycyclic aromatic hydrocarbons (PAHs) were reviewed as the major risk factors for lung cancer development. In this proposal, the investigators collected fifteen kinds of major PAHs and the investigators would like to perform the following studies:

1. Study the gene expression and subcellular localization of GNMT in the normal-tumor tissue pairs of lung cancer patients.
2. Study the associations of the polymorphisms of GNMT in lung cancer patients and the susceptibility to lung cancer;
3. To assess the allelic loss at GNMT and determined the LOH rate of GNMT in the normal-tumor tissue pairs of lung cancer patients.
4. Study the associations of the copy number variation (CNV) of GNMT and the susceptibility to lung cancer;
5. Study the interaction between GNMT and polycyclic aromatic hydrocarbons (PAHs) in lung cancer cell lines.

DETAILED DESCRIPTION:
Multi-functional protein Glycine N-methyltransferase (GNMT, EC2.1.1.20, localized to chromosome 6p12), affects genetic stability by a) regulating the ratio of S-adenosylmethionine (SAM) to S-adenosylhomocystine (SAH) and b) binding to folate. Based on the following observations, GNMT is classified as a tumor susceptibility gene: a) diminished GNMT expression levels in both human hepatocellular carcinoma (HCC) cell lines and tissues; b) genotypic analyses of several human GNMT gene polymorphisms showed a loss of heterozygosity in 36-47% of the genetic markers in HCC tissues and also related to the susceptibility of prostate cancer; c) GNMT binds to environmental carcinogens such as benzo(a)pyrene (BaP) and aflatoxin B1 (AFB1) and protect the liver cells by inhibiting DNA-adduct formation.

Environmental carcinogens such as polycyclic aromatic hydrocarbons (PAHs) were reviewed as the major risk factors for lung cancer development. In this proposal, the investigators collected fifteen kinds of major PAHs and would like to perform the following studies:

1. Study the gene expression and subcellular localization of GNMT in the normal-tumor tissue pairs of lung cancer patients.
2. Study the associations of the polymorphisms of GNMT in lung cancer patients and the susceptibility to lung cancer;
3. To assess the allelic loss at GNMT and determined the LOH rate of GNMT in the normal-tumor tissue pairs of lung cancer patients.
4. Study the associations of the copy number variation (CNV) of GNMT and the susceptibility to lung cancer;
5. Study the interaction between GNMT and polycyclic aromatic hydrocarbons (PAHs) in lung cancer cell lines.

So far, the investigators have analyzed the gene expression of GNMT in the normal-tumor tissue pairs of some lung cancer patients. The investigators also analyzed the interaction between the GNMT and some PAHs using lung cancer cell lines. These data are helpful to clarify the susceptibility of lung cancer patients with the gene expression in GNMT.

This study is helpful in elucidating the role of GNMT plays in the tumorigenesis of lung cancer which may have important implications in the development of strategies for the prevention, diagnosis and treatment of lung cancer and other types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a lung cancer patient.

Exclusion Criteria:

* Participant is under 18 years old.
* Participant is not a lung cancer patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-10